CLINICAL TRIAL: NCT02725671
Title: Cardiogoniometry for Detecting Coronary Artery Disease by CT Angiography
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor enrollment due to insufficient study support.
Sponsor: Johns Hopkins University (Other)
Collaborators: Enverdis Corp. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB00033908
Record Dates: First submitted 2016-03-10; First posted 2016-04-01 (Estimated); Results first posted 2020-02-25 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2020-06

CONDITIONS: Coronary Heart Disease; Coronary Artery Disease; Ischemic Heart Disease
MeSH Terms: conditions — Coronary Disease; Coronary Artery Disease; Myocardial Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cardiogoniometry and ECG Assessment (Other): The same patient will undergo both advanced ECG assessment using cardiogoniometry and standard ECG
  Interventions: Device: Explorer

INTERVENTIONS:
Device: Explorer — ECG device which records comprehensive voltage potential data in the myocardium

SUMMARY:
Cardiogoniometry is a technique to process and evaluate vectorcardiography from regular ECG acquisitions. Vectorcardiography has a long tradition in cardiology for providing comprehensive information on myocardial function and integrity. In recent years, computer assisted analysis has allowed automated interpretation of vectorcardiography with promising results in comparison to standard ECG for identifying patients with coronary heart disease. This study aims to investigate the utility of cardiogoniometry for noninvasively identifying patients who are at risk from coronary heart disease.

DETAILED DESCRIPTION:
Cardiogoniometry is a technique to process and evaluate vectorcardiography from regular ECG acquisitions. Vectorcardiography has a long tradition in cardiology for providing comprehensive information on myocardial function and integrity. Compared to standard electrocardiography, vectorcardiography has shown to be more sensitive to detect structural and ischemic heart disease. Unfortunately, the interpretation of vectorcardiography is complex which has hindered its widespread application. In recent years, computer assisted analysis has allowed automated interpretation of vectorcardiography with promising results in comparison to standard ECG for identifying patients with ischemic heart disease. However, the underlying mechanisms and threshold of altered cardiac vectors in the presence of coronary artery disease are not well understood. This research aims at exploring the relationship of computer assisted analysis of vectorcardiography with the presence, extent, severity, and location of coronary artery disease in comparison to standard ECG evaluation. Furthermore, the investigators intent to follow up enrolled patients for the occurrence of adverse cardiovascular events for correlation with test findings. These data will provide comprehensive information on the diagnostic performance of noninvasive, inexpensive evaluation of cardiac vector loops for identifying patients at risk from coronary artery disease. Specifically, the study aims to:

1. Compare the diagnostic accuracy of cardiogoniometry with standard ECG for detecting coronary artery disease as assessed by CT angiography
2. Investigate the relationship between abnormal cardiogoniometry findings and the extent/severity/location of coronary artery disease by CT angiography
3. Compare the intermediate term prognosis of patients according to cardiogoniometry, standard ECG, and CT findings

ELIGIBILITY:
Inclusion Criteria:

* Patients age 18 or older who are referred for elective cardiac CT examination for evaluation of coronary artery disease

Exclusion Criteria:

* hemodynamic instability
* history of anaphylactic contrast reaction
* inability of following breath hold instructions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2015-04; Primary Completion 2019-04 (Actual); Study Completion 2020-06-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Armin A Zadeh, MD PhD MPH, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Study Group: Single study group. All patients are planned to undergo both tests, Cardiogoniometry (CGM) and CT angiography.
Period: Overall Study
Arm/Group | Study Group
Started | 2
Completed | 1
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Groups:
- Study Group: Single study group. All patients are planned to undergo both tests, CGM and CT angiography.
Arm/Group | Study Group
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 1
Age, Continuous [Mean (Full Range); unit: years] | 56 [44 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2
Cardiac Risk Factors [Count of Participants; unit: Participants] — Number of patients with traditional risk factors, i.e., Hypertension, Diabetes Mellitus, Hyperlipidemia, smoking will be recorded.
  Participants | 2

OUTCOME MEASURES:

1. Primary Outcome: Accuracy of Identifying Patients With at Least One 50 Percent or Greater Coronary Artery Stenosis by CT Angiography
Description: Area under curve (AUC) analysis is proposed to be used to determine the diagnostic accuracy of cardiogoniometry for detecting patients with coronary heart disease as defined by at least one 50% or greater stenosis on CT coronary angiography.
Time Frame: 30 days from CGM analysis
Population: Minimum data needed for this measure was not collected and therefore could not be calculated.
Arm/Group | Study Group
Number analyzed (Participants) | 0

2. Secondary Outcome: Accuracy of Identifying Patients With Any Coronary Atherosclerotic Disease by CT Angiography
Description: Area under the curve (AUC) analysis is proposed to be used to asses the diagnostic accuracy of CGM for identifying patients with any coronary atherosclerotic disease
Time Frame: 30 days
Population: Insufficient enrollment for analysis for this outcome measure
Arm/Group | Study Group
Number analyzed (Participants) | 0

3. Secondary Outcome: Incidence of Death at Follow up
Description: Patient follow up data will be used to performance of CGM to identify patients who are at risk of suffering adverse cardiac events at follow up compared to coronary CT angiography using AUC analysis.
Time Frame: 5 years after enrollment
Population: Insufficient enrollment for analysis of this outcome measure
Arm/Group | Study Group
Number analyzed (Participants) | 0

4. Secondary Outcome: Risk of Myocardial Infarction
Description: Incidence of myocardial infarction at follow up
Time Frame: 5 years after enrollment
Population: Insufficient enrollment for analysis of this outcome measure
Arm/Group | Cardiogoniometry and ECG Assessment
Number analyzed (Participants) | 0

5. Secondary Outcome: Risk of Revascularization at Follow up
Description: Incidence of revascularization at follow up
Time Frame: 5 year after enrollment
Population: Insufficient enrollment for analysis of this outcome measure
Arm/Group | Cardiogoniometry and ECG Assessment
Number analyzed (Participants) | 0

6. Secondary Outcome: Risk of Hospitalization
Description: Incidence of hospitalization at follow up
Time Frame: 5 years after enrollment
Population: Insufficient enrollment for analysis of this outcome measure
Arm/Group | Cardiogoniometry and ECG Assessment
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 4 years
Arm/Group | Cardiogoniometry and ECG Assessment
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-04-03): https://cdn.clinicaltrials.gov/large-docs/71/NCT02725671/Prot_SAP_000.pdf